CLINICAL TRIAL: NCT06492694
Title: Evaluation of a Fish Oil-based, Essential-oil Infused Supplement on Markers of Health
Brief Title: Omega-3 Supplement and Health Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dōTERRA International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DO-124023-OWO
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Fish oil; Omega-3; Gene expression; Wild orange essential oil
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oil + wild orange essential oil supplement (Experimental): Participants in this arm will take three capsules of a fish oil + wild orange essential oil supplement daily for approximately six weeks.
  Interventions: Dietary Supplement: Fish oil + wild orange essential oil supplement
- Fish oil supplement (Active Comparator): Participants in this arm will take three capsules of a fish oil essential oil supplement daily for approximately six weeks.
  Interventions: Dietary Supplement: Fish oil supplement

INTERVENTIONS:
Dietary Supplement: Fish oil + wild orange essential oil supplement — This supplement contains fish oil and wild orange essential oil as its active ingredients.
  Arms: Fish oil + wild orange essential oil supplement
Dietary Supplement: Fish oil supplement — This supplement contains fish oil as its active ingredient.
  Arms: Fish oil supplement

SUMMARY:
The goal of this clinical trial is to learn whether fish oil-based supplements can affect gene expression and serum protein markers in healthy volunteers. The main questions it aims to answer are:

1. How does daily ingestion of fish oil supplements affect gene expression, omega-3 levels, and protein markers as measured in blood?
2. How does daily ingestion of fish oil supplements affect anthropometric measurements?
3. How does daily ingestion of fish oil supplements affect subjective quality of life and health parameters?
4. Do fish oil + wild orange essential oil supplements produce different outcomes than fish oil supplements alone?
5. Is ingesting fish oil supplements daily safe, as measured by laboratory tests and adverse events?

Researchers will compare two types of fish oil supplements. One type contains fish oil and wild orange essential oil as its active ingredients. The other type contains only fish oil as its active ingredient.

Participants will:

* Be assigned one of the two types of fish oil supplements
* Take three softgels of their assigned supplement every day for about six weeks
* Attend two study visits in which they provide blood and urine samples, complete subjective health and quality of life assessments, and undergo anthropometric measurements
* Complete weekly subjective health assessments from home

DETAILED DESCRIPTION:
This randomized, double-blind study will recruit healthy adults to compare gene expression profile, omega-3 levels, and protein markers before and after consumption of fish oil supplements for approximately six weeks. Quality of life will also be assessed using subjective surveys and questionnaires. Safety markers (liver and kidney function, hematology, urinalysis, and adverse events) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-64 years old

  * Local to Pleasant Grove, Utah, and/or willing to come to the clinical research center for study visits
  * Willing to provide blood and urine samples during study visits
  * Willing and able to consume study product daily for about 6 weeks
  * Willing to track consumption of study product
  * Willing to keep diet, exercise, sleeping, and current non-study supplement use the same throughout the study
  * Willing to avoid alcohol, recreational drugs, and smoking/vaping for the duration of the study (approximately 7 weeks)
  * Willing to wash out of all internally-consumed essential oil and botanical products for at least 2 weeks prior to starting the study and willing to maintain the washout for the duration of the study (about 9 weeks)
  * Willing to receive and respond to regular texts, emails, and/or phone calls from study staff
  * No metabolic disease (BMI>35, diagnosis and treatment of hypertension, diabetes, or dyslipidemia)
  * No major diseases under treatment by a doctor (Medical Reviewer's discretion)
  * No pregnancy within the last 60 days or currently breastfeeding (females)
  * No allergy to fish oil, olive oil, or orange essential oil
  * No regular internal consumption of orange essential oil within the last 1 month (regularly is defined as dosing daily for more than 2 consecutive weeks, or dosing more than 2-3 times per week for 4 consecutive weeks)
  * No regular internal consumption of omega-3 or other fish oil supplements within the last 1 month (regularly is defined as dosing daily for more than 2 consecutive weeks, or dosing more than 2-3 times per week for 4 consecutive weeks)
  * No alcohol, recreational drug, or smoking/vaping use in the past 1 month
  * No evidence of medical condition, significant disease or disorder, medication, or surgery within the past 12 months that may, in the judgment of the medical provider, put the participant at risk or affect study results, procedures, or outcomes
  * Not currently or previously participating in any other clinical trial within the last 30 calendar days
  * Signed informed consent, HIPAA Authorization, and Confidentiality Agreement

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Gene expression | 6 weeks
  Gene expression analysis refers to a genome-wide quantification of methylation. EPIC850k array will be used for methylation analysis. This represents approximately 900,000 gene locations. The main feature performed is a differential methylation analysis to determine what has significantly changed from one time point to another.
Interleukin 6 (pg/mL) | 6 weeks
  Serum marker for inflammation
High sensitivity C-reactive protein (mg/L) | 6 weeks
  Serum marker for inflammation and cardiac health
Apolipoprotein B (mg/dL) | 6 weeks
  Serum marker for cardiovascular disease risk
Total cholesterol (mg/dL) | 6 weeks
  Item in lipid panel for efficacy assessment
Triglycerides (mg/dL) | 6 weeks
  Item in lipid panel for efficacy assessment
High density lipoprotein (HDL) Cholesterol (mg/dL) | 6 weeks
  Item in lipid panel for efficacy assessment
Very Low density lipoprotein (VLDL) Cholesterol (mg/dL) | 6 weeks
  Item in lipid panel for efficacy assessment
Low density lipoprotein (LDL) Cholesterol (mg/dL) | 6 weeks
  Item in lipid panel for efficacy assessment
Omega-3 blood levels (%) | 6 weeks
  Assessment of omega-3 fatty acid concentration in blood

SECONDARY OUTCOMES:
Albumin (g/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Blood urea nitrogen (BUN) (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Creatinine (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Alkaline phosphatase (U/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Alanine transaminase (ALT) (U/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Aspartate aminotransferase (AST) (U/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Calcium (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Carbon Dioxide (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Chloride (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Potassium (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Sodium (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Total bilirubin (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Total protein (g/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Body mass index (BMI) | 6 weeks
  Determine whether body mass index is affected by the consumption of the study product.
Blood pressure (mmHg) | 6 weeks
  Determine whether blood pressure is affected by the consumption of the study product.
Heart rate (BPM) | 6 weeks
  Determine whether heart rate is affected by the consumption of the study product.
White blood cells (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Red blood cells (x10E6/uL) | 6 weeks
  Item in complete blood count for safety assessment
Hemoglobin (g/dL) | 6 weeks
  Item in complete blood count for safety assessment
Hematocrit (%) | 6 weeks
  Item in complete blood count for safety assessment
Mean corpuscular volume (fL) | 6 weeks
  Item in complete blood count for safety assessment
Mean corpuscular hemoglobin (pg) | 6 weeks
  Item in complete blood count for safety assessment
Mean corpuscular hemoglobin concentration (g/dL) | 6 weeks
  Item in complete blood count for safety assessment
Red cell distribution width (%) | 6 weeks
  Item in complete blood count for safety assessment
Platelets (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Neutrophils (%) | 6 weeks
  Item in complete blood count for safety assessment
Lymphocytes (%) | 6 weeks
  Item in complete blood count for safety assessment
Monocytes (%) | 6 weeks
  Item in complete blood count for safety assessment
Eosinophils (%) | 6 weeks
  Item in complete blood count for safety assessment
Basophils (%) | 6 weeks
  Item in complete blood count for safety assessment
Neutrophils (Absolute) (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Lymphocytes (Absolute) (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Monocytes (Absolute) (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Basophils (Absolute) (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Immature granulocytes (%) | 6 weeks
  Item in complete blood count for safety assessment
Immature granulocytes (Absolute) (x10E3/uL) | 6 weeks
  Item in complete blood count for safety assessment
Safety/tolerability | 6 weeks
  This study will monitor the occurrence and frequency of adverse events and safety, both through participant report and blood chemistry/hematology analyses.
Generalized Anxiety Disorder-7 (GAD-7) scale | 6 weeks
  Self-reported scale for the measurement of anxiety severity
Patient Health Questionnaire (PHQ-8) scale | 6 weeks
  Self-reported scale for the measurement of depression severity
Leeds Sleep Evaluation Questionnaire (LSEQ) scale | 6 weeks
  Self-reported scale for the measurement of sleep quality
Short Form-20 (SF-20) scale | 6 weeks
  Self-reported scale for assessment of subjective quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stevens, PhD, Principal Investigator — doTERRA International
Locations (1):
- doTERRA International, Pleasant Grove, Utah, United States